CLINICAL TRIAL: NCT00175227
Title: Prevention of Contrast-Induced Nephropathy: a Randomized Controlled Trial of Saline + Furosemide + Mannitol in High Risk Patients Undergoing Cardiac Angiography
Brief Title: Prevention of Contrast-Induced Nephropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Heritage Foundation for Medical Research (Other)
Responsible Party: Sumit Majumdar/Principal Investigator, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HSRIF #96-20
Record Dates: First submitted 2005-09-10; First posted 2005-09-15 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-05

CONDITIONS: Contrast-induced Nephropathy; Acute Renal Failure; Chronic Renal Failure
Keywords: contrast-induced nephropathy; prevention; renal failure; cardiac angiogram
MeSH Terms: conditions — Acute Kidney Injury; Kidney Failure, Chronic; Renal Insufficiency | interventions — Mannitol; Furosemide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Saline hydration + mannitol + furosemide
  Interventions: Drug: intravenous saline hydration + mannitol + furosemide
- Controls (Placebo Comparator): Saline hydration without mannitol or furosemide
  Interventions: Drug: intravenous saline hydration

INTERVENTIONS:
Drug: intravenous saline hydration + mannitol + furosemide — 500 mls half-normal saline + 25g mannitol + 100 mg furosemide
  Arms: Intervention
Drug: intravenous saline hydration — 500 mls half-normal saline
  Arms: Controls

SUMMARY:
Patients with pre-existing kidney disease are at high risk of acute renal failure when exposed to radio-contrast dyes, for example during a cardiac angiogram.

The investigators hypothesize that an infusion of saline + furosemide + mannitol will reduce rates of contrast-induced nephropathy when compared with saline infusion controls.

DETAILED DESCRIPTION:
Patients with pre-existing kidney disease are at high risk of acute renal failure when exposed to radio-contrast dyes, for example during a cardiac angiogram.

We hypothesize that an infusion of saline + furosemide + mannitol will reduce rates of contrast-induced nephropathy when compared with saline infusion controls.

We define an episode of contrast nephropathy using the conventional often published definition of a 25% relative increase in serum creatinine OR a 44 umol absolute increase in serum creatinine within 48 hours of contrast exposure.

ELIGIBILITY:
Inclusion Criteria:

* age > 21 years
* serum creatinine > 150 umol/L
* able and willing to provide informed consent

Exclusion Criteria:

* known hypersensitivity to contrast, furosemide, or mannitol
* unable to tolerate a fluid load (e.g., acute pulmonary edema)
* ESRD, on dialysis
* previous enrollment in this study or previous contrast administration with the last 2 weeks
* refusal by treating physician

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 1996-05; Primary Completion 2000-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients that develop contrast-induced nephropathy after cardiac angiography | Within 48 hours of angiogram

SECONDARY OUTCOMES:
Safety of the intervention based on transfer to ICU, need for dialysis, or death | During hospitalization episode
Adverse clinical events and measures of renal function | 6 weeks post-angiogram
Health related quality of life | 6 weeks post-angiogram
Subgroup analyses based on (a) diabetes; (b) amount of contrast; and (c) baseline creatinine | Within 48 hours of angiogram

CONTACTS AND LOCATIONS:
Overall Officials: Sumit R Majumdar, MD, MPH, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospitals, Edmonton, Alberta, Canada

REFERENCES:
- [Result] Majumdar SR, Kjellstrand CM, Tymchak WJ, Hervas-Malo M, Taylor DA, Teo KK. Forced euvolemic diuresis with mannitol and furosemide for prevention of contrast-induced nephropathy in patients with CKD undergoing coronary angiography: a randomized controlled trial. Am J Kidney Dis. 2009 Oct;54(4):602-9. doi: 10.1053/j.ajkd.2009.03.024. Epub 2009 Jun 17. PMID 19535188
- [Derived] Hashimoto H, Yamada H, Murata M, Watanabe N. Diuretics for preventing and treating acute kidney injury. Cochrane Database Syst Rev. 2025 Jan 29;1(1):CD014937. doi: 10.1002/14651858.CD014937.pub2. PMID 39878152